CLINICAL TRIAL: NCT03115905
Title: A Registry Study for Emergency Medical Service of Aneurysmal Subarachnoid Hemorrhage With Different Economic Development Levels Areas in China
Brief Title: A Registry Study for Emergency Medical Service of Aneurysmal Subarachnoid Hemorrhage in China
Acronym: CIAP-5
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Hongqi Zhang, MD, chairman of the neurosurgery department of Xuanwu hospital, Xuanwu Hospital, Beijing
Other Study IDs: 2016YFC1300805
Record Dates: First submitted 2017-03-29; First posted 2017-04-14 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Emergency Medical Services
Keywords: Aneurysmal Subarachnoid Hemorrhage; Emergency Medical Services; Registry Study; China
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a staged registry study of early treatment strategy management of acute aneurysmal subarachnoid hemorrhage(aSAH) among different economic development levels areas in China.

First stage, the study will investigate and register the basic information of emergency treatment management for the acute aSAH in 20 different grade centers located in different economic levels districts including Northeast part, Northern, Eastern, South-central, Northwest, Southwest and Qinghai-Tibet of China. Comparing the the outcome of acute aSAH to find the critical factors to affect it by statistical analysis. Then,the investigators will offer some suggestions to adjust the measures to improve the efficacy of emergency medical service for acute SAH.

Second stage, to evaluate the outcome after applying the new suggestion of self-control methods.

The investigators hypothesis that there is an appropriate green pathway in different districts to shorten the rescuing time, improve the curative effects.

DETAILED DESCRIPTION:
For this study, the investigators consulted and hired professionals and experts about data collection, data analysis and methodology. So it has an intact systematic Project Steering Committee for the whole project, including Data Monitoring Committee, Data Management Committee, Project Academic Committee, Executive Group, Project Manager, Project Statistician,Technical Support Center. Also the project have a scientific regulations system.

Steering Committee: To monitor and supervise the progress of the Registry Study for Emergency Medical Service of Aneurysmal Subarachnoid Hemorrhage With Different Economic Development Levels Areas in China toward its interim and overall objectives.To consider recommendations of the data monitoring committee and local ethics committees. To promote the publicity and presentation of all aspects of this trial.

Project Manager and Executive Group: To ensure the successfully implementation of this project, including charging the daily operations of the study in 20 different research hospitals, organizing the monthly meeting to consider issues raised during the monthly progress of the study, liaising with the steering committee,the data management centre and statistical centre.

Data management Committee: To be responsible for setting up and maintain the Electronic Data Capture (EDC) System according to the paper Case Report Form(pCRF) designed by principal investigators. To collect and save the pCRF coming from sub-centers. To entry the data into EDC system and keep the same with CRF. To organize training for the investigators about the rules in filling the EDC and pCRF.To determine the frequency of the Data Management Report and to fed it back to the steering committee every three months.

Data Monitoring Committee: To determine the frequency of the data monitoring including the source data(Medical records) accuracy, completeness and representativeness comparing the external data(EDC, pCRF) in 20 centers. To report the results after the monitoring back to the steering committee about the missing data, non-reported and other problems about the study. To make a Standard Operation Procedure(SOP) from getting data to using data.

Academic Committee: To supervise the academic issues including patient recruitment, protocol deviation, adverse events evaluating. To settle down the question and problem in the process of the study.

Project Statistician: The investigators cooperate with the statisticians of Medical Research & Biometrics Center National Center for Cardiovascular Diseases, China to get the professional statistical report.

Technical Support Center: To provide technical support during the process of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Proven subarachnoid haemorrhage on computed tomography(CT) or lumbar puncture less than 14 days.
2. Exist at least one target intracranial aneurysm demonstrated by computed tomography angiography (CTA) or Digital Subtraction Angiography(DSA).
3. Age is older than 14 years old.
4. Patient or relatives agreed to sign the consent form.

Exclusion Criteria:

1. Some special types of controversial aneurysmal subarachnoid hemorrhage such as caused by blood blister-like aneurysm,dissection aneurysm and so on.
2. Participation in another randomised drug or clinical trial for subarachnoid hemorrhage.
3. Refusal of consent.
4. Women during pregnancy.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who diagnosed as aneurysmal subarachnoid hemorrhage in emergency.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
the rate of modified Rankin Score(mRS) higher than 3. | 3 months after treatment
  It means that the rate of disability and mortality.

OTHER OUTCOMES:
The rate of treatment success | Immediate evaluating after treatment
  We defined the aneurysm was totally or nearly occluded identified by the Digital Subtraction Angiography(DSA).
The rate of treatment success | Six months after treatment.
  We defined the aneurysm was totally or nearly occluded identified by the Digital Subtraction Angiography(DSA).
The rate of main adverse events | duration of hospital stay
  We defined the main adverse events includes any deaths and ischemia or hemorrhage related to the treatment during 30 days after treatment, and neurologic complications from 30 days after treatment to 1 year.
The rate of main adverse events | 3 months after discharge.
  We defined the main adverse events includes any deaths and ischemia or hemorrhage related to the treatment during 30 days after treatment, and neurologic complications from 30 days after treatment to 1 year.
The rate of main adverse events | 6 months after discharge.
  We defined the main adverse events includes any deaths and ischemia or hemorrhage related to the treatment during 30 days after treatment, and neurologic complications from 30 days after treatment to 1 year.
The rate of main adverse events | 1 year after discharge.
  We defined the main adverse events includes any deaths and ischemia or hemorrhage related to the treatment during 30 days after treatment, and neurologic complications from 30 days after treatment to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Zhang, PhD. M.D, Principal Investigator — Xuanwu hosptial,Capital Medical University,China
Locations (2):
- China (2):
  - Beijing Neurosurgical Institute, Beijing, Beijing Municipality
  - Neurosurgery Department of Xuanwu hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
we can share the original data 5 years after the study.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: THE DATA WILL BE SHARED IN 2024 AND LAST FOR EVER.
Access Criteria: SEND EMAIL TO SISSI.CCMU@FOX.COM AND STATE THE PURPOSE AND USE.

REFERENCES:
- [Result] Molyneux A, Kerr R; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group; Stratton I, Sandercock P, Clarke M, Shrimpton J, Holman R. International Subarachnoid Aneurysm Trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomized trial. J Stroke Cerebrovasc Dis. 2002 Nov-Dec;11(6):304-14. doi: 10.1053/jscd.2002.130390. PMID 17903891
- [Result] Darsaut TE, Raymond J. Barrow Ruptured Aneurysm Trial: 3-year results. J Neurosurg. 2013 Dec;119(6):1642-4. doi: 10.3171/2013.5.JNS13917. Epub 2013 Aug 30. No abstract available. PMID 23991842
- [Result] Thomas AJ, Ogilvy CS. ISAT: equipoise in treatment of ruptured cerebral aneurysms? Lancet. 2015 Feb 21;385(9969):666-8. doi: 10.1016/S0140-6736(14)61736-0. Epub 2014 Oct 28. No abstract available. PMID 25465112
- [Result] Molyneux AJ, Birks J, Clarke A, Sneade M, Kerr RS. The durability of endovascular coiling versus neurosurgical clipping of ruptured cerebral aneurysms: 18 year follow-up of the UK cohort of the International Subarachnoid Aneurysm Trial (ISAT). Lancet. 2015 Feb 21;385(9969):691-7. doi: 10.1016/S0140-6736(14)60975-2. Epub 2014 Oct 28. PMID 25465111
- [Result] Mitha AP, Ogilvy CS. ISAT: coiling or clipping for ruptured intracranial aneurysms? Lancet Neurol. 2005 Dec;4(12):791-2. doi: 10.1016/S1474-4422(05)70231-3. No abstract available. PMID 16297834
- [Result] Britz GW. ISAT trial: coiling or clipping for intracranial aneurysms? Lancet. 2005 Sep 3-9;366(9488):783-5. doi: 10.1016/S0140-6736(05)67190-5. No abstract available. PMID 16139637
- [Derived] Hou X, Geng J, Wang S, Fan X, Xiang S, Hu P, He C, Li M, Zhang H. High-resolution magnetic resonance imaging (HRMRI) for judging the location of paraclinoid aneurysms (PAs): assisting in diagnosis and treatment decision of PAs. Chin Neurosurg J. 2026 Jan 26;12(1):3. doi: 10.1186/s41016-025-00420-8. PMID 41588479
- [Derived] Guo X, Guo F, Xuan L, Zhang X, He C, Zhang H, Zhang T. Short-Term Extreme Temperatures, Temperature Fluctuations, and the Risk of Aneurysmal Subarachnoid Hemorrhage: A Nationwide Case-Crossover Study. Stroke. 2026 Jan;57(1):134-147. doi: 10.1161/STROKEAHA.125.052300. Epub 2025 Nov 7. PMID 41200812